CLINICAL TRIAL: NCT04070677
Title: Prospective, Multicenter Clinical Study Assessing the Effect of ZIVEREL® on the Symptomatic Treatment of Radiation Oesophagitis in Cancer Patients
Brief Title: Clinical Study Assessing the Effect of ZIVEREL® in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Collaborators: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ZESRAD
Record Dates: First submitted 2019-06-26; First posted 2019-08-28 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Acute Esophagitis
Keywords: Acute Esophagitis; Radiotherapy; Ziverel; Chondroitin sulfate; Hyaluronic acid; Poloxamer 407; Chemoradiotherapy; Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ziverel arm (Experimental): Patients included will receive treatment with ZIVEREL®, initially 10 mL every 8 hours, 30 minutes after meals, to avoid physical entrainment by food, during a minimum of 8 weeks, recruited during a period of 12 months. The treatment will be indicated when the patient develops a radiation-induced esophagitis of degree ≥ 2.
  Interventions: Combination Product: Ziverel

INTERVENTIONS:
Combination Product: Ziverel — Patients in treatments with radiotherapy alone (RT) or radiochemotherapy (RT-CH) with acute radiation-induced esophagitis grade 2 or superior according to the most recent CTCAE will received support treatment with ZIVEREL®

SUMMARY:
Radiation-induced esophagitis is an acute, dose-limiting toxicity in oncologic treatment. Since it can lead to interruption of treatment, hospitalization, and even death, clinicians should be aware of this condition as an adverse effect of oncologic therapies, in order to prevent interruption of treatment, as it has been associated with reduced survival. ZIVEREL® is a new, over-the-counter medical device that comes as an oral solution in a 10-ml stick pack. It is composed of hyaluronic acid, chondroitin sulfate, and poloxamer 407 and Women plays a role in the symptomatic relief of esophagitis induced by radiotherapy alone or radiochemotherapy in oncologic patients. ZIVEREL® acts naturally and exerts a protective action by reinforcing the effect of the elements that make up the extracellular matrix, where the connective tissue provides the architecture, proteoglycans maintain the fluid-electrolyte balance, and glycoproteins maintain the intracellular substrate responsible for cell-cell reactions and cell-matrix reactions. The objective of this study is to evaluate whether administration of ZIVEREL® diminishes the grade of acute radiation-induced esophagitis and the incidence of severe esophagitis in oncologic patients treated with radiotherapy or radiochemotherapy.

DETAILED DESCRIPTION:
Hyaluronic acid is a glycosaminoglycan formed by glucuronic acid and N acetylglucosamine disaccharide units. It is found mainly in the extracellular matrix of the loose connective tissue and is associated with several key processes, including cell signaling and repair, as well as with tissue generation, morphogenesis, and structural organization of the extracellular matrix itself. In clinical terms, its role is well known in conditions such as mouth ulcers, where its barrier effect relieves symptoms. Chondroitin sulfate forms part of the glycosaminoglycan group in the extracellular matrix, which is in turn formed by D-glucuronic acid and N-acetylgalactosamine. It has been shown to protect the epithelium of the esophageal mucosa by shielding the epithelial areas damaged by acid, thus diminishing catabolic activity and inhibiting proteolytic enzymes (e.g., metalloproteases, collagenase, or elastase). Chondroitin sulfate also regulates several inflammatory mediators (TNF-α, IL-1β, COX-2, PGE2, and NFκB) and reduces the synthesis of nitric oxide, which is involved in the inflammatory cascade. Polaxamer 407 is a bioadhesive component that acquires the active ingredients of ZIVEREL® adhere to the damaged mucosa and are not dragged away by the ingestion of food and liquids.

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS 0-1.
* Signature of informed consent.
* Patients with any type of neoplasm that requires treatment with radiotherapy or radiochemotherapy, and who develop a radiation-induced esophagitis of degree ≥ 2 (according to CTCAE v4.03)
* Hematological function (neutrophils ≥2000 / ml, platelets ≥100000 / ml, hemoglobin> gr / dl), hepatic (bilirubin <1.5) and renal acceptable (glomerular filtration rate> 50 ml / min).
* Patients without contraindication for the administration of ZIVEREL®, in accordance with the instructions for use of the product.

Exclusion Criteria:

* ECOGPS≥2
* Hypersensitivity for some of the active ingredients or a component of ZIVEREL®
* Alteration in haematological function (neutrophils ≤2000 / ml, platelets ≤100000 / ml, hemoglobin <8gr/dl), hepatic (bilirubin> 1.5) and/or glomerular filtration rate <50 ml/min).
* Patients who have a medical history of psychiatric disorders or any other condition that interfere with the study
* Patients with esophageal candidiasis or oral cavity candidiasis at the time of entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Symptomatic relief of radiation-induced esophagitis grade ≥2 in cancer patients undergoing radiotherapy and radiochemotherapy after administration of ZIVEREL®. | 1 year
  Symptomatic relief of radiation-induced esophagitis grade ≥2

SECONDARY OUTCOMES:
Dosimetric prognostic factors | 1 year
  Determine the dosimetric prognostic factors in the development of radiation induced esophagitis (Dmed, Dmax, V5, V15, V20, V30, V35, V40, V45, V50, V60)
Analyze the health-related quality of life during the treatment | 1 year
  EORTC QLQ-C30 (version 3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No